CLINICAL TRIAL: NCT01637285
Title: A Phase 1, Randomized, Open-label, Parallel-group Study To Evaluate The Pharmacokinetics Of Pf-04856883 (Cvx-096) Following Subcutaneous Administration In Healthy Volunteers
Brief Title: A Pharmacokinetic Study of CVX-096 (PF-04856883) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: B1111005
Record Dates: First submitted 2012-06-26; First posted 2012-07-11 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-04856883 Treatment Arm 1 (Experimental)
  Interventions: Biological: PF-04856883
- PF-04856883 Treatment Arm 2 (Experimental)
  Interventions: Biological: PF-04856883
- PF-04856883 Treatment Arm 3 (Experimental)
  Interventions: Biological: PF-04856883
- PF-04856883 Treatment Arm 4 (Experimental)
  Interventions: Biological: PF-04856883

INTERVENTIONS:
Biological: PF-04856883 — Dose A
  Arms: PF-04856883 Treatment Arm 1
Biological: PF-04856883 — Dose B
  Arms: PF-04856883 Treatment Arm 2
Biological: PF-04856883 — Dose C
  Arms: PF-04856883 Treatment Arm 3
Biological: PF-04856883 — Dose D
  Arms: PF-04856883 Treatment Arm 4

SUMMARY:
The purpose of the study is to further evaluate the PK characteristics of PF-04856883.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
PF-04856883 Pharmacokinetics including Cmax, Tmax, AUCo-infinity, AUClast, Cl/F, Vz/F and t1/2 | 4 weeks

SECONDARY OUTCOMES:
Number of subjects with AEs reported | 4 weeks
Number of subjects with abnormal physical examination findings | 4 weeks
Number of subjects with abnormal clinical laboratory results | 4 weeks
Number of subjects with abnormal ECGs | 4 weeks
Number of subjects with abnormal vital signs | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States